CLINICAL TRIAL: NCT05438706
Title: A Clinical Study of the Efficacy and Safety of Chidamide in Combination With Camrelizumab and Carboplatin or Capecitabine in the Second and Third Line Treatment of Relapsed/Metastatic Triple-negative Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xichun Hu, MD, Fudan University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSIIT-C21
Record Dates: First submitted 2022-06-25; First posted 2022-06-30 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Triple-negative Breast Cancer
Keywords: chidamide; camrelizumab; carboplatin; capecitabine; relapsed/metastatic; triple-negative breast cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Neoplasm Metastasis | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; camrelizumab; Carboplatin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): chidamide in combination with camrelizumab and capecitabine
  Interventions: Drug: chidamide; Drug: camrelizumab; Drug: capecitabine
- Arm 2 (Experimental): chidamide in combination with camrelizumab and carboplatin
  Interventions: Drug: chidamide; Drug: camrelizumab; Drug: carboplatin

INTERVENTIONS:
Drug: chidamide — Chidamide, an HDAC inhibitor
Drug: camrelizumab — Camrelizumab (AiRuiKa™), a programmed cell death 1 (PD-1) inhibitor being developed by Jiangsu Hengrui Medicine Co. Ltd, recently received conditional approval in China for the treatment of relapsed or refractory classical Hodgkin lymphoma. The drug is also being investigated as a treatment for various other malignancies, including B cell lymphoma, oesophageal squamous cell carcinoma, gastric/gastroesophageal junction cancer, hepatocellular carcinoma, nasopharyngeal cancer and non-squamous, non-small cell lung cancer.
Drug: carboplatin — Carboplatin [diammine(1,1-cyclobutanedicarboxylato)platinum(II)] is one of the most promising second generation platinum compounds. Its greater chemical stability in comparison with cisplatin accounts for its lower reactivity with nucleophilic sites of DNA.
  Arms: Arm 2
Drug: capecitabine — Capecitabine is an oral prodrug of 5-fluorouracil (5-FU) and approved for treatment of various malignancies. Hereditary genetic variants may affect a drug's pharmacokinetics or pharmacodynamics and account for differences in treatment response and adverse events among patients.
  Arms: Arm 1

SUMMARY:
To evaluate the efficacy and safety of chidamide in combination with camrelizumab and carboplatin or capecitabine in the second and third line treatment of relapsed/metastatic triple-negative breast cancer

DETAILED DESCRIPTION:
This study is a prospective, single-center, single-arm, open-label clinical study. Successfully screened patients with relapsed/metastatic triple-negative breast cancer will receive chidamide and camrelizumab at the prescribed doses Combined with carboplatin or capecitabine therapy, Chidamide single drug should be taken for lead-in therapy before combined therapy.

ELIGIBILITY:
Inclusion Criteria:

1. The patients voluntarily participated in the study and signed the informed consent form
2. 18-75 years old, female
3. EC0G score 0-1
4. Expected survival time ≥ 3 months
5. Patients with recurrent / metastatic breast cancer confirmed by histopathology, with negative expression of ER or PR and negative expression of HER2; Patients with local recurrence need to be confirmed by the investigator that radical resection is impossible
6. Previous anti-tumor regulations (Patients has previously received first-line chemotherapy and disease progression, and at most has received second-line treatment (recurrence and metastasis during adjuvant treatment will be regarded as first-line treatment), Patients who have previously received taxoids drugs)
7. Patients were preferentially enrolled into the chidamide in combination with camrelizumab and capecitabine group( except fo who had failed to receive capecitabine treatment in the past)
8. If the investigator thinks who is suitable to be enrolled in the chidamide in combination with camrelizumab and carboplatin group (such as genetic recombination deficiency, high HRD evaluation score or BRCA1/2 gene mutation, etc.), is preferred to enter this group
9. At least one extracranial measurable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria version 1.1.
10. The functions of important organs meet the following requirements (no blood components and cell growth factors have been used within 2 weeks before enrollment) ANC ≥ 1.5 × 109 /L; PLT ≥ 75 × 109 /L. Hb ≥ 90 g/L TBIL ≤ 1.5×ULN (upper limit of normal) ALT and AST ≤ 2.5×ULN. Urea / urea nitrogen (BUN) and creatinine (CR) ≤ 1.5 × ULN, or creatinine clearance ≥ 60ml/min/1.73m2 Left ventricular ejection fraction (LVEF) ≥ 50% QTcF(Fridericia correction) < 470 ms INR≤1.5×ULN，APTT≤1.5×ULN

Exclusion Criteria:

1. Previously treated with histone deacetylase inhibitors (HDACi)
2. Previously treated with pd-1/pd-l1 inhibitors
3. Untreated imaging confirmed central nervous system metastasis (except asymptomatic brain metastasis)
4. Patients who have received systematic, radical brain or meningeal metastasis treatment (radiotherapy or surgery) in the past, but have been stable for at least 4 weeks as confirmed by imaging, have stopped systemic hormone treatment for more than 2 weeks, and have no clinical symptoms can be included
5. There were ascites, pleural effusion and pericardial effusion with clinical symptoms in the baseline period, requiring drainage, or serous effusion drainage within 4 weeks before the first dose
6. Inability to swallow, intestinal obstruction or other factors affecting drug administration and absorption
7. Systematic treatment such as chemotherapy, molecular targeted therapy or other clinical trial drugs were received within 4 weeks before enrollment, except for observational studies
8. Prior malignancy active within the previous 5 years (except for curable cancers, such as or Non-Melanocytic Tumors of the Skin or carcinoma in situ of the cervix)
9. Had major surgical operation or obvious trauma within 4 weeks before enrollment, or it is expected that the patient will receive major surgical treatment
10. Allergy to the drug components of this study
11. Active HBV and HCV infection; Except for the patients with stable hepatitis B (DNA titer shall not be higher than 500 IU/ml or copy number <1000 copies/ml) and cured hepatitis C (HCV RNA detection is negative)
12. History of immunodeficiency, including HIV test positive, or suffer from other acquired or congenital immunodeficiency diseases, or have a history of organ transplantation
13. Any heart disease, including (1) angina pectoris; (2) Arrhythmia requiring medication or clinically significant; (3) Myocardial infarction; (4) Heart failure; (5) Any other heart disease judged by the researcher as unsuitable for the test; The severity of abnormal cardiac or renal function in screening period is ≥ II
14. Pregnant women, lactating women or fertile women , Or subjects of childbearing age who are unwilling to take effective contraceptive measures during the study period and at least 3 months after the last dose
15. According to the judgment of the investigator, there are concomitant diseases that seriously endanger the safety of the patient or affect the completion of the study (such as severe hypertension, diabetes, thyroid disease, active infection, etc.)
16. History of neurological or mental disorders, including epilepsy or dementia
17. The investigator determined who was not suitable for the study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 70 (Estimated)
Dates: Start 2022-07-10 (Estimated); Primary Completion 2023-11-10 (Estimated); Study Completion 2024-07-10 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | Up to approximately 12 weeks
  ORR is the percentage of participants with the best overall response of complete response (CR) or partial response (PR) according to RECIST 1.1. CR = Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm; PR = At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | Up to approximately 30 months
  PFS defined as the time from the date of randomization to the first evidence of disease progression as defined by response evaluation criteria in solid tumors (RECIST) v1.1 or death from any cause. Progressive Disease (PD) was at least a 20% increase in the sum of the diameters of target lesions, with reference being the smallest sum on study and an absolute increase of at least 5 mm, or unequivocal progression of non-target lesions, or 1 or more new lesions. If a participant does not have a complete baseline disease assessment, then the PFS time was censored at the date of randomization, regardless of whether or not objectively determined disease progression or death has been observed for the participant. If a participant was not known to have died or have objective progression as of the data inclusion cutoff date for the analysis, the PFS time was censored at the last adequate tumor assessment date.
Overall Survival (OS) | Up to approximately 30 months]
  Time from date of randomization to the date of death from any cause
Disease control rate(DCR) | Up to approximately 12 weeks
  DCR is defined as cases where objective remission(assessed as complete remission or partial remission according RECIST 1.1 standard) or stable disease during the study.
Clinical Benefit Rate (CBR) | Up to approximately 12 weeks
  Percentage of participants with complete response (CR) or partial response (PR) or stable disease (SD) lasting 24 weeks or longer as defined in RECIST 1.1.CR = Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm; PR = At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters; SD = Neither sufficient shrinkage to qualify for PR or CR nor an increase in lesions which would qualify for progressive disease: PD = At least a 20% increase in the sum of diameter of all measured target lesions, taking as reference the smallest sum of diameter of all target lesions recorded at or after baseline. In addition to the relative increase of 20% the sum must also demonstrate an absolute increase of at least 5 mm

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided